CLINICAL TRIAL: NCT06051500
Title: Psychological and Physiological Effects of Different Objects of Breath Meditation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 2023-0749; Protocol Version 06/28/2023 (Other: UW Madison); L&S/CTR FOR HEALTHY MINDS (Other: UW Madison)
Record Dates: First submitted 2023-09-11; First posted 2023-09-25 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Physiological Stress; Psychological Stress; Emotions
Keywords: meditation; focus; attention; breath
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Intervention Model Description: Random allocation to one of two sequence of meditation practice.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nostril focus followed by belly focus (Experimental): Participants will be randomly assigned to concentrate on the nostrils first, then the belly second following a period of rest.
  Interventions: Behavioral: Nostril focus followed by belly focus
- Belly focus followed by nostril focus (Experimental): Participants will be randomly assigned to concentrate on the belly first, then the nostrils second following a period of rest.
  Interventions: Behavioral: Belly focus followed by nostril focus

INTERVENTIONS:
Behavioral: Nostril focus followed by belly focus — Focused breathing on the nostrils followed by focus breathing on the belly.
  Arms: Nostril focus followed by belly focus
Behavioral: Belly focus followed by nostril focus — Focused breathing on the bellyfollowed by focus breathing on the nostrils.
  Arms: Belly focus followed by nostril focus

SUMMARY:
The goal of this research is to test whether certain areas of focus in breath meditation are connected with certain mental health outcomes. The main question to be addressed is whether attention placed on the breath in the belly versus the nostrils during meditation results in differences in subjective experience, respiration and heart rate.

Participants will:

* complete surveys
* have heart rate and respiration measured
* practice focused breathing

Participants can expect the study visit to last for one hour.

DETAILED DESCRIPTION:
An online prescreen will determine eligibility. Participants that 1) are under 18, 2) are not students currently enrolled at UW-Madison 3) have previous mediation experience 4) obtain a high PROMIS depression or anxiety score, or 5) have been diagnosed with one or more psychiatric disorders by a healthcare professional that will be listed in the pre-screen survey will be excluded.

Participants deemed eligible following prescreen will schedule a lab visit. At the beginning of the lab visit, participants will be provided a consent document and time to ask questions. After signing the consent form, researchers will place ECG leads and a respiration belt on participants, and then complete the baseline survey battery. Participants will then sit at rest for 5 minutes of baseline heart rate and respiration data collection. Next, participants will be randomly assigned in a counterbalanced order to nostril focus first or belly focus first and asked to follow a brief (~5 minute) guided practice. After the practice, participants will complete a second battery of self-reports and then have a 10-minute period of rest/recovery. They will then complete the second practice (~5 minutes) followed by a final survey. The entire session will take about an hour.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* student at UW Madison
* no major history of meditation practice

Exclusion Criteria:

* under 18 years of age
* not currently enrolled at UW Madison
* have previous meditation experience
* Self-reports a mental health diagnosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2023-10-20 (Actual); Primary Completion 2024-05-02 (Actual); Study Completion 2024-05-02 (Actual)

PRIMARY OUTCOMES:
Change in Positive and Negative Affect Schedule (PANAS-SF) | At baseline; after meditation 1 (5 minutes); and, after meditation 2 (15 minutes)
  PANAS-SF is a 20-item questionnaire to assess positive versus negative affect. 10 of the items indicate positive affect, 10 indicate negative. Scores can range between 10-50 for positive affect, with higher scores representing higher levels of positive affect. Scores can range between 10-50 for negative affect, with lower scores representing lower levels of negative affect.
Change in Respiration | Baseline to practice 1 epoch (10 minutes); baseline 2 to practice 2 epoch (25minutes)
  Using respiration belts, rate of respiration will be collected. Paired with heart rate, this will give us further insight into the physiological responses to the participant's experience of the two variations of breath meditation.
Change in Heart Rate | Baseline to practice 1 epoch (10 minutes); baseline 2 to practice 2 epoch (25minutes)
  Using ECG electrodes and a BIOPAC system, heart rate will be monitored. Paired with respiration rate, this will give us further insight into the physiological responses to the participant's experience of the two variations of breath meditation.

SECONDARY OUTCOMES:
Perseverative Thinking (PTQ) | Baseline only
  The PTQ is a 15-item questionnaire asking how participants typically think about negative experiences or problems. Scores can range from 0-60, with higher scores representing higher levels of perseverative thinking.
Change in Interoceptive Awareness | At baseline; after meditation 1 (5 minutes); and, after meditation 2 (15 minutes)
  The Multidimensional Assessment of Interoceptive Awareness (MAIA) is a 37-item questionnaire that measures multiple dimensions of self-awareness. The Noticing, Attention Regulation and Self-regulation scales will be used. Scores range between from 0-20, 0-35 and 0-20, respectively, with higher scores represent higher interoceptive awareness.
Change in Mindfulness | At baseline; after meditation 1 (5 minutes); and, after meditation 2 (15 minutes)
  The Five Facet Mindfulness Questionnaire (FFMQ) is a 39-item questionnaire. The Non-react to inner experience and Act with awareness subscales will be used. Scores can range from 7-35 and 8-40, respectively; higher scores represent higher levels of mindfulness facet.
Change in Relaxation | At baseline; after meditation 1 (5 minutes); and, after meditation 2 (15 minutes)
  A research assistant or I will ask each participant to respond to the following statement: "In this moment I feel relaxed." Participants will select one of the following responses: strongly disagree, slightly disagree, neither agree nor disagree, slightly agree, strongly agree.
Change in Focus | At baseline; after meditation 1 (5 minutes); and, after meditation 2 (15 minutes)
  A research assistant or I will ask each participant to respond to the following statement: "In this moment I feel focused." Participants will select one of the following responses: strongly disagree, slightly disagree, neither agree nor disagree, slightly agree, strongly agree.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Hirshberg, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
After de-identification, all processed study data will be posted to support open science practices. Heart rate and respiration indices will be posted after processing (i.e., not raw data).